CLINICAL TRIAL: NCT06969261
Title: Adapting the Penny Chatbot for Perinatal OUD Patients: COPILOT
Acronym: PENNY-COPILOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 853729; R34DA058461 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-05-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Perinatal Opioid Use Disorder; Opioid Use Disorder
Keywords: Maternal Health; Maternal Substance Use; Perinatal OUD; Chatbot; mHealth Interventions; Loneliness
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chatbot Intervention (Experimental): This is a single arm study designed to assess the acceptability and feasibility of the chatbot.
  Interventions: Behavioral: Penny COPILOT

INTERVENTIONS:
Behavioral: Penny COPILOT — The Penny COPILOT chatbot is an interactive short messaging system (SMS) program that provides educational and supportive content for postpartum individuals. The chatbot has been adapted to include information relevant to opioid use disorder recovery in order to decrease the risk of returning to use among people who use drugs. Messages are sent at specified intervals relevant to the postpartum course and the chatbot allows for two way messaging with an interactive lens.

SUMMARY:
To address both loneliness and engagement in perinatal and OUD care among perinatal women, the investigators plan to adapt an existing texting support chatbot, Penny, to make it appropriate for use by women who are pregnant and postpartum and dealing with OUD. The newly adapted chatbot, Penny COPILOT, will allow for two way short message service (SMS) messaging to respond appropriately and accurately to user generated input. The investigative team, in collaboration with the Penn Mixed Methods Research Lab (MMRL) and Penn's Way 2 Health Team, will use intervention mapping guided by the Consolidated Framework for Implementation Science. The investigators will conduct a needs assessment, assemble an advisory board, engage in pretesting to ensure safety and refine content, and pilot test the resultant adapted Penny COPILOT in a sample of 20 perinatal women with OUD to evaluate acceptability, feasibility, and patient satisfaction. The goal is to develop and refine an acceptable, feasible, and satisfactory supportive texting chatbot to promote patient engagement in perinatal and OUD care and decrease perceived loneliness.

ELIGIBILITY:
Inclusion Criteria:

* Biological females who are currently pregnant or within 6 weeks postpartum.
* Able to read, write, and speak English at a 6th grade level.
* Diagnosed and receiving treatment for, or willing to receive treatment for opioid use disorder.
* Receiving prenatal care and OUD care at a Penn affiliated hospital.

Exclusion Criteria:

-Current untreated psychosis, mania, or active suicidality as assessed by the Mini International Neuropsychiatric Interview (MINI).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
UCLA Loneliness Scale. | During Aim 3 activities, assessments will occur at Baseline and at 3-month Follow-up.
  The UCLA Loneliness Scale (Version 3) is the most commonly used measure of loneliness, with strong test-retest reliability, high internal consistency, and validity.97 While the word "lonely" is never used explicitly in the 20-item scale, subjects are asked to report the frequency of specific experiences (e.g., "How often do you feel in tune with others around you?") on a 4-point Likert scale (1 = "I never feel this way" to 4 = "I often feel this way.") For dichotomous analysis of loneliness, we will use the loneliness severity threshold adapted from Doryab98 which defines "lonely" as having a score greater than 40, while "not lonely" is defined as having a score less than or equal to 40.

SECONDARY OUTCOMES:
Opioid use questionnaire | During Aim 3 activities, assessments will occur at Baseline and 3-month Follow-up.
  A questionnaire designed by our investigative team that queries a participant's opioid use, specifically identifying their drug of choice, method of administration, pattern of use, triggers for use, frequency and amount of use, barriers to relapse, and recency of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Sara L Kornfield, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified demographic data and responses to survey items will be shared by appropriate request to the study PI.